CLINICAL TRIAL: NCT04672252
Title: The Use of Cannabidiol (CBD) in Pain Reduction and Opioid Use After Shoulder Arthroscopy; A Double-Blind, Randomized Control Study
Brief Title: The Use of Cannabidiol (CBD) in Pain Reduction and Opioid Use After Shoulder Arthroscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Orcosa Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01293
Record Dates: First submitted 2020-11-23; First posted 2020-12-17 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - CBD (Experimental)
  Interventions: Drug: CBD Oral Disintegrating Tablet (ODT)
- Cohort 2 - Placebo (Placebo Comparator)
  Interventions: Other: Placebo ODT

INTERVENTIONS:
Drug: CBD Oral Disintegrating Tablet (ODT) — Cohort 1: CBD ODTs to be administered with routine post-operative pain management regimen
  Arms: Cohort 1 - CBD
Other: Placebo ODT — Cohort 2 will not receive CBD; but a visually indistinguishable placebo ODT instead.
  The resident physician, physician assistant, anesthesiologist, surgeon and study team members will remain blinded. Additionally, all patients will receive a traditional upper extremity interscalene block as per routine.
  Arms: Cohort 2 - Placebo

SUMMARY:
This study is designed to evaluate the effects of administering CBD to control post-operative pain in patients undergoing shoulder arthroscopy. Secondly, the purpose will be to evaluate the effectiveness of CBD in comparison with opioid therapy for post-operative pain.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing an arthroscopic shoulder procedure (rotator cuff repair, decompression, labrum repair)
* Patients ages 18-75, inclusive
* Female patients must be currently practicing effective forms of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (less than 1% per year) when used consistently and correctly
* Male patients must be using an effective form of contraception

Exclusion Criteria

* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Older than 75 years of age
* Any patient considered a vulnerable subject: pregnant women or fetuses, children, cognitively impaired adults, prisoners
* History of cannabis abuse or dependence
* History of coagulation abnormalities and thromboembolic disease or current abnormal coagulation test values
* History of stroke or acute coronary syndromes within 3 months before surgery
* Abnormal coagulation profile
* Renal failure (serum creatinine > 250 μmol/L [2.83 mg/dL]) or liver cirrhosis
* Patients with a history of hypersensitivity to Percocet
* Patients that have been on pre-operative opioid management for any reason
* Patients meeting the DSM-V for major psychiatric illness, such as bipolar disorder
* Patients diagnosed with major depression, psychosis, or substance abuse disorder
* Patients with current or a history of suicidal ideation
* Breastfeeding females
* Patients with clinically significant illness, including cardiovascular disorders
* Clinically significant lab abnormalities
* Abnormal LFTs
* Patients with major neurological disorders, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain/head injury, or seizures
* Patients with moderate (Child-Pugh B) and severe hepatic impairment (Child-Pugh C).
* Patients taking moderate or strong inhibitors of CYP3A4 and CYP2C19 (listed below) concomitantly
* Patients taking strong CYP3A4 and CYP2C19 inducers (listed below) concomitantly
* Patients taking substrates of UTG1A9, UTGB17, CYP2A1, CYP2B6, CYP2C8, CYP2C9 and CYP2C19 (listed below) concomitantly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alaia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Alaia MJ, Li ZI, Chalem I, Hurley ET, Vasavada K, Gonzalez-Lomas G, Rokito AS, Jazrawi LM, Kaplan K. Cannabidiol for Postoperative Pain Control After Arthroscopic Rotator Cuff Repair Demonstrates No Deficits in Patient-Reported Outcomes Versus Placebo: 1-Year Follow-up of a Randomized Controlled Trial. Orthop J Sports Med. 2024 Feb 5;12(2):23259671231222265. doi: 10.1177/23259671231222265. eCollection 2024 Feb. PMID 38322981
- [Derived] Alaia MJ, Hurley ET, Vasavada K, Markus DH, Britton B, Gonzalez-Lomas G, Rokito AS, Jazrawi LM, Kaplan K. Buccally Absorbed Cannabidiol Shows Significantly Superior Pain Control and Improved Satisfaction Immediately After Arthroscopic Rotator Cuff Repair: A Placebo-Controlled, Double-Blinded, Randomized Trial. Am J Sports Med. 2022 Sep;50(11):3056-3063. doi: 10.1177/03635465221109573. Epub 2022 Jul 29. PMID 35905305

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Started | 53 | 47
Completed | 52 | 47
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo | Total
Number analyzed (Participants) | 52 | 47 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.8) | 57.1 (10.1) | 57.65 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 52 | 47 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 52 | 47 | 99
Region of Enrollment [Number; unit: participants]
  United States | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analog Scale (VAS) Score
Description: Pain severity scores at rest will be assessed by use of a visual analog scale (VAS; 0 = no pain, 10 = worst pain imaginable).
Time Frame: Hour 24 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 4.4 (3.1) | 5.7 (3.2)

2. Primary Outcome: Pain Visual Analog Scale (VAS) Score
Description: as for outcome 1
Time Frame: Day 2 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 4.7 (2.8) | 5.3 (2.6)

3. Primary Outcome: Pain Visual Analog Scale (VAS) Score
Description: as for outcome 1
Time Frame: Day 7 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 2.5 (1.9) | 3.2 (2.7)

4. Primary Outcome: Pain Visual Analog Scale (VAS) Score
Description: as for outcome 1
Time Frame: Day 14 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 1.6 (1.4) | 2.3 (2.4)

5. Primary Outcome: Nausea Score on VAS Scale
Description: Any nausea experienced by the patients will be recorded by use of a VAS (0 = no nausea, 10 = worst nausea imaginable).
Time Frame: Day 2 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 2.1 (2.6) | 2.5 (3.1)

6. Primary Outcome: Nausea Score on VAS Scale
Description: Any nausea experienced by the patients will be recorded by use of a VAS (0 = no nausea, 10 = worst nausea imaginable).
Time Frame: Day 7 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 0.2 (1.1) | 0.6 (2.1)

7. Primary Outcome: Nausea Score on VAS Scale
Description: Any nausea experienced by the patients will be recorded by use of a VAS (0 = no nausea, 10 = worst nausea imaginable).
Time Frame: Day 14 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 0.1 (0.4) | 0.5 (1.7)

8. Secondary Outcome: Total Opioid Consumption
Description: Consumption based on patient-self-report
Time Frame: Day 1 Post-Surgery
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
morphine milligram equivalent (MME) | 15.2 (12) | 19.7 (13.6)

9. Secondary Outcome: Total Opioid Consumption
Description: Consumption based on patient-self-report.
Time Frame: Day 2 Post-Surgery
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
morphine milligram equivalent (MME) | 10.3 (18.7) | 16.7 (36.6)

10. Secondary Outcome: Total Opioid Consumption
Description: Consumption based on patient-self-report.
Time Frame: Day 7 Post-Surgery
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
morphine milligram equivalent (MME) | 59.3 (53.2) | 67.3 (55.2)

11. Secondary Outcome: Total Opioid Consumption
Description: Consumption based on patient-self-report.
Time Frame: Day 14 Post-Surgery
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
morphine milligram equivalent (MME) | 8 (19.3) | 10.3 (22.7)

12. Secondary Outcome: Number of Completed Doses Out of 3 Maximum Doses/Day
Description: Based on patient-self-report.
Time Frame: Day 1 Post-Surgery
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
Doses | 2.9 (0.27) | 3 (0)

13. Secondary Outcome: Number of Completed Doses Out of 3 Maximum Doses/Day
Description: Based on patient-self-report.
Time Frame: Day 7 Post-Surgery
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
Doses | 3 (0) | 2.7 (0.95)

14. Secondary Outcome: Number of Completed Doses Out of 3 Maximum Doses/Day
Description: Based on patient-self-report.
Time Frame: Day 14 Post-Surgery
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
Doses | 2.8 (0.4) | 2.7 (1)

15. Secondary Outcome: Patient Satisfaction Score
Description: Patients will record their satisfaction with their management, on a 0-10 scale (where 0= not at all satisfied; and 10 = completely satisfied).
Time Frame: Hour 24 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 7 (3) | 5.6 (3.7)

16. Secondary Outcome: Patient Satisfaction Score
Description: as for outcome 15
Time Frame: Day 2 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 7.3 (2.5) | 6 (3.3)

17. Secondary Outcome: Patient Satisfaction Score
Description: as for outcome 15
Time Frame: Day 7 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 8 (2.6) | 7.9 (2.7)

18. Secondary Outcome: Patient Satisfaction Score
Description: as for outcome 15
Time Frame: Day 14 Post-Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
Number analyzed (Participants) | 52 | 47
score on a scale | 8.7 (2.3) | 8.5 (2.4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Regular laboratory testing for elevated liver enzymes and self-reporting by participants.
Arm/Group | Cohort 1 - CBD | Cohort 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/47
Other Adverse Events (participants affected / at risk) | 4/52 | 4/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - CBD (N=52) | Cohort 2 - Placebo (N=47)
Elevated alanine transaminase (Hepatobiliary disorders) | 4 | 4 — Elevated alanine transaminase at Day 7. All resolved postoperatively by Day 14.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT04672252/Prot_SAP_000.pdf